CLINICAL TRIAL: NCT04103931
Title: Pilot Randomized Trial of a Patient Decision Aid for Treatment of Aortic Stenosis
Brief Title: Impact of a Patient Decision Aid for Treatment of Aortic Stenosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: University of Colorado, Denver (Other)
Responsible Party: Principal Investigator, Karen Sepucha, Associate Professor, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2017P001883
Record Dates: First submitted 2019-09-24; First posted 2019-09-26 (Actual); Last update posted 2022-01-05 (Actual); Status verified 2021-12

CONDITIONS: Aortic Valve Stenosis
Keywords: Shared Decision Making
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Intervention Model Description: Patients are randomly assigned to receive the decision aid or usual care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): Participants will receive usual care and will not get the decision aid to review.
- Patient Decision Aid (Experimental): Participants in this arm will receive the patient decision aid, titled "Treatment Choices for Aortic Stenosis" to review.
  Interventions: Behavioral: "Treatment Choices for Aortic Stenosis" Decision Aid

INTERVENTIONS:
Behavioral: "Treatment Choices for Aortic Stenosis" Decision Aid — A decision aid, titled "Treatment Choices for Aortic Stenosis," produced by the American College of Cardiology that contains information for patients deciding between TAVR and surgery to treat their aortic stenosis.
  Arms: Patient Decision Aid

SUMMARY:
This project will evaluate the impact of a patient decision aid created by the American College of Cardiology for patients considering treatment of aortic stenosis. The decision aid describes surgical aortic valve replacement (SAVR) surgery and transcatheter valve replacement surgery (TAVR).

DETAILED DESCRIPTION:
The pilot trial will enroll patients who are coming in to see a valve specialist (cardiac surgeon or interventional cardiologist) to discuss treatment options for aortic stenosis. The study will recruit patients at Massachusetts General Hospital or at the University of Colorado Health Heart and Vascular Center, Anschutz Medical in Denver, Colorado and randomly assign them to usual care arm or decision aid arm. The decision aid will be given to the participant in clinic at the time of their appointment. Patient participants in both arms will be asked to complete a short survey after the visit. The survey will assess knowledge, treatment preference, shared decision making (SDM), and decisional conflict. Analyses will compare the two arms on these outcomes to generate preliminary data on impact of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18-85 years only
* English speaking
* Severe aortic stenosis, defined as an aortic valve area < 1 cm2
* Never had AVR or who had previous AVR > 6 months previous
* Patients perceived by the clinician to be at low or intermediate risk for SAVR

Exclusion Criteria:

* Concomitant disease of another heart valve or the aorta that required either transcatheter or surgical intervention

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2019-09-23 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Knowledge score | About 1 week after receiving the decision aid
  Patients will complete 6 multiple choice knowledge items and a total knowledge score (0-100%) will be created by summing the number of correct responses and dividing by the number of items.

SECONDARY OUTCOMES:
Shared Decision Making Process score | About 1 week after receiving the decision aid
  Items from the SDM Process survey will be summed to create a total score (0-4) with higher scores indicating more shared decision making.
Treatment Preference | About 1 week after receiving the decision aid
  Patients will indicate their preferred treatment (TAVR, surgery, or unsure)
Treatment received | 12-21 weeks post visit
  Chart review will determine type of treatment received (e.g. TAVR, SAVR, other)

OTHER OUTCOMES:
SURE scale | About 1 week after receiving the decision aid
  The 4 item SURE scale will measure decisional conflict and the percent with the top score (4 out of 4) will be reported
CollaboRATE scale | About 1 week after the visit
  The 3 item Collaborate scale will be scored and the percent receiving the top score (27 out of 27) will be reported

CONTACTS AND LOCATIONS:
Overall Officials: Karen R Sepucha, PhD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - University of Colorado Denver I Anschutz Medical Campus, Aurora, Colorado
  - Massachusetts General Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The study team will create a complete, cleaned, de-identified copy of the final data set.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: The data will be made available to outside investigators starting 6 months after publication.
Access Criteria: Information about the data sets will be on the Health Decision Sciences Center website and in publications of the data. Dr. Sepucha will share a de-identified data set with outside investigators at no cost, according to approved Massachusetts General Hospital (MGH)/ Mass General Brigham policies for data sharing. Investigators from other sites will be able to request the data and will be required to complete a data use agreement that ensures that all local Institutional Review Board (IRB) requirements are met before using the data, that they will not attempt to identify any data in the dataset, and that they will not share the data set with anyone outside their project team.